CLINICAL TRIAL: NCT02744833
Title: A Randomized Phase I/II Study to Assess the Safety, Tolerability, and Efficacy of GMI-1271 in Patients With Calf-Level Deep Venous Thrombosis
Brief Title: Study to Assess Safety, Tolerability, and Efficacy of GMI-1271 in Patients With Calf-level Deep Venous Thrombosis (DVT)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The trial was funded in part by a grant; the trial closed when the grant ended.
Sponsor: GlycoMimetics Incorporated (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMI-1271-220
Record Dates: First submitted 2016-04-08; First posted 2016-04-20 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Deep Venous Thrombosis
Keywords: DVT
MeSH Terms: conditions — Venous Thrombosis | interventions — uproleselan; enoxaparin sodium; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GMI-1271 (Experimental)
  Interventions: Drug: GMI-1271
- Enoxaparin Sodium (Lovenox®) (Active Comparator)
  Interventions: Drug: Enoxaparin Sodium (Lovenox®)

INTERVENTIONS:
Drug: GMI-1271
  Arms: GMI-1271
Drug: Enoxaparin Sodium (Lovenox®)
  Arms: Enoxaparin Sodium (Lovenox®)

SUMMARY:
This study will evaluate the safety profile of GMI-1271 and its effect on thrombus resolution in patients with distal calf vein Deep Venous Thrombosis (DVT).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Male or female
* Diagnosed with acute isolated calf vein Deep Venous Thrombosis (DVT)
* Willing and able to participate in all required evaluations and procedures in this study protocol

Exclusion Criteria:

* History or presence of clinically significant medical condition or disease in the opinion of the principal investigator
* Uncontrolled acute life-threatening bacterial, viral or fungal infection
* Unable to be treated with systemic anticoagulants
* Current use of immunosuppressants, antiplatelets (other than aspirin), anticoagulants, and/or anti-epileptics
* Diagnosis of acute leukemia or multiple myeloma undergoing active treatment or maintenance treatment within the past 5 years
* Current or recent cancer treatment
* Major surgery within 21 days or planned surgery during the study period
* Female subjects who are pregnant or breastfeeding
* Known history of HIV, Hepatitis B or Hepatitis C
* Alcoholism or drug use
* Clinically significant cardiovascular disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of GMI-1271 in patients with calf-level DVT by assessment with vital signs, standard laboratory blood tests, electrocardiogram, and adverse event evaluation. | 19 days
  Adverse events will be assessed via Common Terminology Criteria for Adverse Events (CTCAE 4.03).

SECONDARY OUTCOMES:
To evaluate the effects of GMI-1271 on thrombus resolution or stabilization as measured by Doppler ultrasound | 19 days
To evaluate the effects of GMI-1271 on the incidence of bleeding time | 19 days
To evaluate the effects of GMI-1271 on bleeding markers such as Prothrombin time (PT) | 19 days
To evaluate the effects of GMI-1271 on biomarkers of coagulation | 19 days

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sood, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States